CLINICAL TRIAL: NCT01801943
Title: Walking Interventions, Cognitive Remediation and Mild Cognitive Impairment
Acronym: WalkCog-MCI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: participants are no longer being examined or receiving intervention
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PBRC 12032
Record Dates: First submitted 2013-02-26; First posted 2013-03-01 (Estimated); Last update posted 2022-09-23 (Actual); Status verified 2014-06

CONDITIONS: Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Population Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cognitive Remediation Therapy Group (Experimental): 30 minute Cognitive Remediation Therapy and 60 minute Healthy Living Class three time per week
  Interventions: Behavioral: Cognitive Remediation Therapy Group
- Walking Intervention Group (Experimental): 60 minutes of walking and 30 minutes of reading stimulation three times a week
  Interventions: Behavioral: Walking Intervention (WI) Group
- Combination Group (Experimental): 30 minutes of Cognitive Remediation therapy and 60 minutes of walking three times a week
  Interventions: Behavioral: Combination Group
- Healthy Living Group (Experimental): 60 minute Healthy Living Class and 30 minutes of reading stimulation three times a week.
  Interventions: Behavioral: Healthy Living Group

INTERVENTIONS:
Behavioral: Cognitive Remediation Therapy Group — 30 min Cognitive Remediation Therapy + 60 Min Healthy Living class 3x week
  Arms: Cognitive Remediation Therapy Group
Behavioral: Walking Intervention (WI) Group — 60 min Walking Intervention + 30 min low interface reading 3x week
  Arms: Walking Intervention Group
Behavioral: Combination Group — 30 min Cognitive Remediation Therapy + 60 min Walking Intervention 3x week
  Arms: Combination Group
Behavioral: Healthy Living Group — 60 Min Healthy Living class + 30 min low interface reading 3x week
  Arms: Healthy Living Group

SUMMARY:
The purpose of this study is to determine the effects of a coordinated intervention of cognitive remediation training (CRT) and walking intervention on cognition and gait in the elderly.

DETAILED DESCRIPTION:
This is a single blind randomized study designed to understand the effects of different interventions, walking interventions and cognitive remediation in particular, towards cognition and gait in the elderly. The study uses a 4 arm approach consisting of 4 intervention groups, with each intervention lasting for 12 weeks. The investigators will investigate the effect of each intervention towards cognitive function and gait. All interventions will be conducted on site at the Pennington Biomedical Research Center, and will be focused on determining the effects of different combinations of walking, cognitive remediation, healthy living courses, and reading. Cognitive measures will include objective clinical measures related to dementia, and the gait analysis will include in clinic and "free living" measures related to falls.

ELIGIBILITY:
Inclusion Criteria:

* Men and women meeting all criteria listed below will be included in the study:
* Subjects between 65-85 years of age inclusive
* Subjects with Short Physical Performance Battery of 10 or greater
* Subjects averaging less than 5,000 steps per day
* Subjects with Mini Mental State Exam 25-28, inclusive
* Subjects with normal for age physical-neurological exam
* Subjects able to walk a city block without a walking aid
* Written Informed Consent obtained PRIOR to performing any study procedures

Exclusion Criteria:

* Subjects with difficult walking due to pain or posture
* Subjects with difficulty in using computer due to significant visual and/or fine motor impairment
* Subjects with large weight loss (>15 Kilogram) in the last 12 months
* Subjects with geriatric depression scale > 9.
* Subjects with Malignancies in the past 5 years, with the exception of skin cancer therapeutically controlled
* Subjects with abnormal electrocardiogram results. These include: a resting heart rate below 40 bpm or above 100 bpm, previously unknown and/or untreated atrial fibrillation or flutter, evidence of a third degree A-V block, a previously undocumented left bundle branch block, S-T segment depression of greater than 2 mm, evidence of a previous MI, or any other findings that in the clinical judgment of the medical investigator preclude participation in an exercise intervention.
* Subjects with shortness of breath, exertional angina, uncontrolled high blood pressure or any other chronic medical condition deemed by the physician to preclude participation in an exercise intervention.
* Subjects with any other medical condition or disease that is life-threatening or that can interfere with, or be aggravated by, exercise.
* Subjects who currently smoke.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Dates: Start 2013-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Effects of interventions on cognition | 6 months
  Standard psychometric tests will be used to measure cognition

SECONDARY OUTCOMES:
Effects of interventions on gait | 6 months
  Standard laboratory assessments and accelerometers will be used to measure gait.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Keller, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States